CLINICAL TRIAL: NCT02593409
Title: HIV Pre-Exposure Prophylaxis Priming of Immune Effectors
Brief Title: HIV PrEP Priming of Immune Effectors
Acronym: PREPPIE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: MRC/UVRI and LSHTM Uganda Research Unit (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PREPPIE001
Record Dates: First submitted 2015-10-21; First posted 2015-11-02 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: HIV-1 Infections
Keywords: HIV-1; pre-exposure prophylaxis (PrEP); immune response
MeSH Terms: interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- TDF/FTC (Other): All participants receive pre-exposure prophylaxis in the form of a daily tablet containing 300 mg of tenofovir disoproxil fumarate and 200 mg emtricitabine (Truvada®, Gilead) for one year, with an optional extension for 6 months.
  Interventions: Drug: TDF/FTC

INTERVENTIONS:
Drug: TDF/FTC — All participants receive pre-exposure prophylaxis in the form of a daily tablet containing 300 mg of tenofovir disoproxil fumarate and 200 mg emtricitabine (Truvada®, Gilead) for one year, with an optional extension for 6 months.
  Other Names: Truvada®

SUMMARY:
Can HIV-specific immunity develop in HIV uninfected humans exposed to HIV whilst receiving antiretroviral pre-exposure prophylaxis (PrEP)? Investigators will investigate this possibility in commercial sex workers in Kampala who will be receiving Truvada PrEP for one year.

DETAILED DESCRIPTION:
Design This will be a single centre open label longitudinal observational trial. Women attending the "Good Health for Women" clinic will be informed about the objectives of the trial and volunteers able to provide informed consent and with high risk of exposure to HIV-1 determined by a sexual history questionnaire will be screened by Rapid antibody test. Seronegatives will be checked for eligibility by clinical examination and laboratory tests. The endpoint for enrolment will be 220 uninfected high risk participants.

Baseline blood samples will be obtained from participants at month 0. A monthly diary card will be provided for self documenting sexual exposure, alcohol use and pill taking. Participants will receive provisions of PrEP (tenofovir disoproxil fumarate (TDF) and emtricitabine (FTC) sufficient for one month, will be instructed on the daily prophylaxis and on how to record adherence on the diary card. Participants will be asked to return each month for treatment re-provisioning and a new card. The content of the diary card will be discussed in a short interview each month.

At month 6 and 12 blood samples will be collected for evaluating immune responses to HIV-1. Additional tests will be done for monitoring HIV-1 status, pregnancy and sexually transmitted infections (STIs). After month 12 PrEP will be discontinued (unless participants opt to continue PrEP until the end of the follow up) and all participants will provide blood samples at month 18.

Baseline and follow-up peripheral blood mononuclear cells (PBMC) samples will be compared for T cell responses to HIV by interferon-γ (IFN-γ) enzyme-linked immunospot (ELISPOT). In case of a positive immune response, plasma collected at the same time point will be nucleic acid test (NAT) tested to verify absence of HIV infection.

HIV infected participants will be evaluated for cluster of differentiation 4 (CD4) T cells and viral load and referred to a Care Program (PEPFAR).

At month 6, 12 and 18 in-depth interviews will be conducted with a randomly selected sample of 44 women (20 percent) to discuss facilitators and barriers to adherence. The diary answers will be tabulated to look for patterns and trends. A framework approach to analysis will be used for the analysis of the qualitative data from interviews.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 at screening
* not intending to move away from the clinic's catchment area for the next 2 years
* HIV-1 antibody negative
* reports commercial sex work
* contact information is provided
* written informed consent

Exclusion Criteria:

* HIV infection at screening
* participation in previous or concurrent HIV vaccine trials
* lactating, pregnant or planning pregnancy
* renal function impairment (serum creatinine >1.5 mg/dl), Fanconi syndrome
* abnormal liver function tests (AST/ALT > 43 U/L), liver disease, viral hepatitis, hepatitis B virus (HBV) infection
* serum phosphorus <2.2mg/dl, osteoporosis
* known sensitivity to components of the Truvada® formulation
* any immunosuppressive treatment, such as systemic corticosteroids
* assumption of medication that interacts with Truvada®
* high likelihood of poor adherence to PREP and clinic attendance
* any condition that in the opinion of the attending physician could endanger the health of the participant or render her unsuitable to participate in the trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2017-05-25 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Change in IFN-γ ELISPOT response to HIV-1 peptides in persistently uninfected individuals between baseline and 12 months on PREP | 0-12 months

SECONDARY OUTCOMES:
Change in IFN-γ ELISPOT response to HIV-1 peptides in persistently uninfected individuals between baseline and 6 months on PREP | 0-6 months
Change in IFN-γ ELISPOT response to HIV-1 peptides in persistently uninfected individuals between 12 months on PREP and at 18 months after PREP cessation | 12-18 months

OTHER OUTCOMES:
HIV-1 incidence. | 0-18 months
Viral load among participants who become infected with HIV-1 despite PREP. | 0-18 months
Adherence to PREP as measured by plasma sampling. | 0-18 months
Adherence to PREP as measured by pill counts. | 0-18 months
Adherence to PREP as measured by participant self-report. | 0-18 months

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Pala, MD, Principal Investigator — MRC/UVRI and LSHTM Uganda Research Unit
Locations (1):
- MRC/UVRI Uganda Research Unit on Aids - Good Health for Women Project, Kampala, Uganda

REFERENCES:
- [Background] Cranage M, Sharpe S, Herrera C, Cope A, Dennis M, Berry N, Ham C, Heeney J, Rezk N, Kashuba A, Anton P, McGowan I, Shattock R. Prevention of SIV rectal transmission and priming of T cell responses in macaques after local pre-exposure application of tenofovir gel. PLoS Med. 2008 Aug 5;5(8):e157; discussion e157. doi: 10.1371/journal.pmed.0050157. PMID 18684007